CLINICAL TRIAL: NCT05184855
Title: Blueberry Supplementation and Inflammation Resolution After Exercise
Brief Title: Blueberries and Exercise Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-0213
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Muscular Injury
Keywords: blueberries; exercise; inflammation; oxylipins; cytokines
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — blueberry extract

STUDY DESIGN:
Intervention Model Description: Randomized, parallel groups
Who Masked: Participant, Investigator
Masking Description: Blueberry powder supplement and a carbohydrate- and fiber-matched placebo powder with flavoring, aroma, and coloring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry (Experimental): 26 g freeze-dried blueberry powder per day or approximately one cup fresh blueberries equivalent; two weeks intake.
  Interventions: Dietary Supplement: Blueberry
- Placebo (Placebo Comparator): 26 g placebo powder per day matched for color, taste, aroma; two weeks intake.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blueberry — Blueberry powder intake
  Arms: Blueberry
Dietary Supplement: Placebo — Placebo powder intake
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if 2-weeks supplementation with blueberries (1 cup/day) compared to placebo can mitigate muscle soreness and damage, and improve inflammation resolution and metabolic recovery during a 5-day period after engaging in an acute, 90-minute bout of eccentric exercise. The primary outcome will be plasma oxylipin levels, extending previously collected data showing that blueberry ingestion decreases post-exercise oxylipins generated from cytochrome P450 enzymes.

DETAILED DESCRIPTION:
Participants will be randomized to the blueberry or placebo groups. The parallel group design is being utilized in this study because of the "repeat exercise bout" effect (i.e., post-exercise muscle damage and inflammation are reduced when the same bout is repeated within days and weeks of the first bout). Participants will come to the lab at 7:00 am at the beginning of the 2-week supplementation period, and then Monday (eccentric exercise bout) and Tuesday through Friday (recovery) in an overnight fasted state. Seven blood samples will be collected and analyzed for various measures of muscle damage, oxylipins, and inflammation. After each of the blood draws, participants will provide a muscle soreness rating (DOMS). Three 24 h urine samples will be collected and analyzed for key metabolic markers of blueberry ingestion.

Visit #1 Pre-Study Study participants will come to the performance lab for orientation to study procedures. This will include a review of the consent form, completion of basic questionnaires, and an introduction to the eccentric muscle exercise bout and the strength/power performance testing protocol (about 1.5 hours) (visit #1). During visit #1, participants will be given two 3-day food records with thorough written and oral instructions on recording procedures (with food models). The 3-day food records will be completed on a Thursday, Friday, and Saturday sequence prior to visits #2 and #3. During visit #1, participants will be given three 24 h urine collection bottles with thorough written and oral instruction on collection procedures. The 24 h urine collection bottles will be collected on the day before visits #2, #3, and #7.

This will be followed by another lab session for pre-study measurements and sample collection (visit #2). Participants will be randomized to blueberry or placebo groups, and provided a 2-weeks supply of supplements. Participants in the blueberry and placebo groups will consume 26 g/d powder mixed in water each day in split doses (half in the morning, half in the afternoon). Compliance will be checked weekly through email correspondence from the Research Manager. A 3-day food record will be collected at the beginning and end of the 2-week supplementation period to assess the background diet. The 3-day food record will be turned in and reviewed by the research team, and analyzed for nutrient and flavonoid content using the Food Processor Version 11.1 (ESHA Research, Salem, OR, USA). ESHA's port utility (Version 4.0; ESHA Research, Salem, OR, USA) will be used to upload the Flavonoid Values for USDA Survey Foods and Beverages (FNDDS) 2007-2010 database. Food/beverage intake will be assessed for macro- and micro-nutrients, total flavonoids and subtotals for each of the six flavonoid subclasses, and three individual flavonoid values (quercetin, cyanidin, and epigallocatechin gallate (EGCG)).

The study will include 5 other lab visits during a one-week period starting on a Monday (visit #3), with morning visits at 7:00 am on Tuesday through Friday (visits 4-7). At each of the 7 lab visits, study participants will come to the lab at 7:00 am not having consumed food or beverages (other than water) for at least the previous 9 hours, and having abstained from vigorous exercise for at least the previous 24-48 hours. The Monday session will take about 2.5 hours (7:00 to 9:30 am), and the Tuesday through Friday sessions will take about 30-45 minutes each. The total amount of time participants will be asked to volunteer for this study is about 8-9 hours at the performance lab.

Baseline Testing (Visit #2) Participants will come to the lab at 7:00 am in an overnight fasted state dressed in exercise clothes. Participants will provide a blood sample using standard phlebotomy procedures. Participants will turn in their 24 h urine collection bottle and 3-day food record. Height, body weight, and body composition will be measured in a private section of the lab. Bioelectrical impedance (BIA) using the seca BIA scale will be used to assess body composition (i.e., the percent of body weight that is fat tissue) and body weight. Participants will remove shoes and socks and stand with bare feet on the seca scale for about 7-10 seconds while using the hands to grasp the side rails. Percent body fat will also be measured using the BodPod. Participants will sit inside the BodPod with a tight-fitting swim suit for about 10 minutes while body fat is calculated. Delayed onset of muscle soreness (DOMS) will be assessed using a 1-10 scale.

Participants will perform some light exercises to warm up, followed by five muscle function tests: vertical jump, bench press, leg-back strength, anaerobic power through the 30-second Wingate test, and 60-yard shuttle run.

1. Vertical jump: Participants will first stand erect with the feet flat on the floor and reach as high as possible with both arms and hands (standing reach height). Participants will then squat down and jump as high as possible with one arm and hand, and tap the measuring device on the Vertec vertical jump apparatus (jump height). This will be repeated three times, with the best score recorded as the difference between the jump and standing reach heights.
2. Bench press to exhaustion at 50%/75%: Participants will lie down supine on a bench, and with spotters standing on either side attempt to bench press a weighted bar equal to 75% (males) or 50% (females) body weight as many times as possible (to a metronome set at 60 beats/min or 30 lifts/min). The bar must touch a foam block on the chest lightly in the down position, and the arms must be straight in the up position.
3. Leg-Back Strength: Leg/lower back strength will be assessed with a dynamometer. With the legs slightly bent at the knee, participants will grasp a bar attached via a chain and a force measuring device with straight arms, and then lift up with maximal effort for several seconds. This will measure the isometric strength of both legs and back, and will be repeated three times.
4. 30-Second Wingate Cycling Test, Anaerobic Power: The Lode cycle ergometer will be adjusted to the participant's body weight (7 watts per kilogram). After a warm up, participants will sprint cycle at maximal speed for 30 seconds. The peak power and average power will be recorded and adjusted to body weight.
5. 60-Yard Shuttle Run Test: The shuttle run is a test of speed and agility. Participants will run back and forth to 5 yards, 10 yards, and 15 yards, for a total of 60 yards. Participants are required to touch the line with their hand at each turn, and run through the finish line. The test involves five touches. The time to complete the test in seconds is recorded. The score is the best time of three trials.

Testing Sequence, Day of Eccentric Muscle Exercise (Monday, Visit #3) and 4-Days Recovery (Tuesday through Friday) (Visits #4-7):

Participants will come to the lab at 7:00 am in an overnight fasted state (i.e., no food or beverages other than water for at least the previous 9 hours). Participants will turn in their 24 h urine collection bottle and 3-day food record. Participants will be weighed and then provide a blood sample, and give a DOMS rating. The blueberry or placebo supplements (half dose) will be consumed mixed in water. Participants will perform some light exercises to warm up, followed by five muscle function tests: vertical jump, bench press, leg-back strength, anaerobic power through the 30-second Wingate test, and shuttle run. Participants will take these performance tests before and after the 90-minute eccentric muscle exercise bout, and each of the following four mornings at the performance lab.

After taking the five performance tests, participants will engage in 90-minutes of eccentric exercise. Immediately following exercise, participants will provide a muscle soreness rating and a blood sample. Participants will then take the five muscle function tests. Participants will ingest the supplements (half dose) during the afternoon (3-6 pm). Participants will return at 7:00 am in an overnight fasted state four days in a row (Tuesday through Friday) after Monday's eccentric exercise bout, and provide DOMS ratings, and blood samples followed by ingestion of the supplements (half dose). Following ingestion of the supplements, participants will take the five muscle function tests. Participants will consume the second half dose of the supplements in the afternoon (Tuesday, Wednesday, Thursday). On Friday morning, participants will provide blood, turn in their 24 h urine sample, and take the supplement (half dose) prior to the muscle function tests. During this week of testing, participants will engage in normal training.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18-50 years.
* Non-smoker.
* Body mass index less than 18.5-30 kg/m2 (not obese).
* Not engaged in regular resistance training (less than 3 sessions per week).
* Agree to train normally, maintain weight, and avoid the regular use of protein supplements, large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation and immune function (especially Advil, Motrin, aspirin, and similar anti-inflammatory drugs) for the duration of the study. (Participant will review supplement and medication use with the Research Manager during orientation).
* Agree to avoid consuming all berries including blueberries, raspberries, and strawberries.
* Agree to consume no more than an average of five servings per day of vegetables and fruit.
* Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis.

Exclusion Criteria:

* Inability to comply with study requirements.
* Engaged in regular resistance training (3 or more sessions per week, on average).
* Body weight below 110 pounds.
* Pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).
* History of allergic reactions to blueberry ingestion.
* Postmenopausal.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of pro-inflammatory oxylipins: 19-hydroxy-eicosatetraenoic acid (HETE), 20-HETE, 20-cooh-AA, 8,9-dihydroxy-eicosatrienoic (all ng/ml) acid; (diHETrE), 14,15-diHETrE | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Inflammation biomarkers

SECONDARY OUTCOMES:
Serum concentration of creatine kinase | Change from pre-exercise to post-exercise (immediately after, and 1-, 2-, 3-, and 4-days after
  Muscle damage biomarker
Urine concentration of hippuric acid | Change from pre-supplementation to post-2-weeks supplementation of blueberries or placebo
  Blueberry metabolite biomarker

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Will provide data upon request.